CLINICAL TRIAL: NCT02136186
Title: Home Telemonitoring in Patients at High Risk for Readmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Brooks Health System (Unknown)
Responsible Party: Principal Investigator, Nancy L. Dawson, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-003548
Record Dates: First submitted 2014-04-16; First posted 2014-05-12 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Inpatients
Keywords: home telemonitoring; readmission; high risk

STUDY DESIGN:
Who Masked: Participant
Masking Description: patients deidentified
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): patients will receive standard of care discharge instructions
- Philips Telehealth (Active Comparator): patients will be discharged with a telemonitoring device for 30 days
  Interventions: Device: Philips Telehealth

INTERVENTIONS:
Device: Philips Telehealth — patients will be provided with a philips home telemonitoring system post hospital discharge
  Arms: Philips Telehealth

SUMMARY:
This study will evaluate the efficacy of home telemonitoring as an intervention to decrease hospital readmissions in patients at high risk for readmission. The overall readmission rate for high-risk MCF hospital patients is approximately 20%. Currently a system is in place to identify and score all MCF patients for their risk of readmission. This score is based on multiple variables including but not limited to: co-morbid conditions, patient's health literacy, whether they are a Medicare/Medicaid patient, their in-home social support, and whether they have had prior hospital admissions within the previous year. The literature shows that home telemonitoring of patients has had mixed results for effectiveness at preventing hospitalizations and emergency department visits. Many of these reports have restricted studies to patients with specific diseases or general characteristics; some have shown improved results while others have not. No study has examined patients who are high risk for readmission to determine if home telemonitoring for 30 days post-discharge reduces the risk for 30-day readmission.

DETAILED DESCRIPTION:
We hope to enroll a total of 1900 participants, 950 in each arm, over the next 2 years. One arm will be the telemonitoring group and one arm will be the standard of care group. Participants will be in the study for 30 days. Participants in the telemonitoring group will receive a Telestation, blood pressure monitor, and pulse oximeter. If the participant also has congestive heart failure, they will receive a scale. All of these vital measurements are to be taken on a daily basis along with survey questions on how the patient feels. If set parameters are out of the normal range, a flag will trigger that requires follow up/intervention from a nurse by telephone. In some cases, the participant might need to come back in to see a physician through the outpatient clinic. The participant in the standard of care group will be contacted via phone 30 days after discharge to learn if they were readmitted to any hospitals or had any emergency room visits during the past 30 days. This data will be collected via Philips software and also entered into the RedCap database here at Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria:

1) readmission risk score of 11 or higher 2) may be from any service in the hospital 3) patient discharged home or 4) patient discharged to skilled nursing/rehabilitation

Exclusion Criteria:

1. international
2. under age 18
3. discharged to hospice
4. discharged to a sub-acute care hospital
5. transferred to an acute care hospital or
6. if the patient has a planned readmission within the next 30 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Readmissions into Hospital | 30 days
  Compare 30-day readmission rates between high-risk patients who are home monitored using technology and high-risk patients who receive the current standard care.

SECONDARY OUTCOMES:
Changes in Readmissions in the Emergency Room | 30 days
  Compare 30-day emergency department visit rates between high-risk patients who are home monitored using technology and high-risk patients who receive current standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Dawson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawson NL, Hull BP, Vijapura P, Dumitrascu AG, Ball CT, Thiemann KM, Maniaci MJ, Burton MC. Home Telemonitoring to Reduce Readmission of High-Risk Patients: a Modified Intention-to-Treat Randomized Clinical Trial. J Gen Intern Med. 2021 Nov;36(11):3395-3401. doi: 10.1007/s11606-020-06589-1. Epub 2021 Jan 27. PMID 33506388
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials